CLINICAL TRIAL: NCT06438094
Title: The Influence of Non-Carious Cervical Lesions on Root Coverage by Means of Coronally Advanced Flap and a Connective Tissue Graft: A Prospective Cohort Study
Brief Title: The Influence of Non-Carious Cervical Lesions on Root Coverage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gonzalo Blasi (Other)
Responsible Party: Sponsor-Investigator, Gonzalo Blasi, Clinical professor, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER-ECL-2022-01
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: There are two treatments but they are based on the tooth-level
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type A gingival recession defects (Experimental): Gingival recession defects that present with a visible CEJ. These defects will receive root coverage surgery only.
  Interventions: Procedure: Root coverage surgery by means of a coronally advanced flap combined with a connective tissue graft
- Type B gingival recession defects (Experimental): Gingival recession defects that do not present a visible CEJ. A cervical composite restoration will be done prior to root coverage surgery.
  Interventions: Procedure: Reconstruction of the CEJ with a composite restoration followed by root coverage surgery by means of a coronally advanced flap combined with a connective tissue graft

INTERVENTIONS:
Procedure: Root coverage surgery by means of a coronally advanced flap combined with a connective tissue graft — A root coverage surgery will be performed using Zucchelli et al.'s coronally advanced flap combined with a connective tissue graft from the palate.
  Arms: Type A gingival recession defects
Procedure: Reconstruction of the CEJ with a composite restoration followed by root coverage surgery by means of a coronally advanced flap combined with a connective tissue graft — Reconstruction of the CEJ with a composite restoration will be performed in B+ and B- defects prior to root coverage surgery. A root coverage surgery will be performed using Zucchelli et al.'s coronally advanced flap combined with a connective tissue graft from the palate.
  Arms: Type B gingival recession defects

SUMMARY:
The goal of this prospective cohort study is to evaluate the effect of non-carious cervical lesions (NCCLs) on the outcome of root coverage therapy. The main question it aims to answer is: In gingival recessions associated with NCCLs, characterized by an undetectable cemento-enamel junction (CEJ), reconstruction of the CEJ with a cervical composite restoration, prior to root coverage surgery by means of a coronally advanced flap combined with a connective tissue graft (CAF+CTG), provides similar clinical and patient-reported outcomes, as compared to the treatment of gingival recessions associated with NCCLs, characterized by a visible CEJ, with root coverage surgery only, by means of a CAF+CTG.

In NCCLs where the CEJ is undetectable (B-type defect), the CEJ will be reconstructed before surgery with a cervical composite restoration mimicking the anatomic features of the contralateral, homologous tooth. CAF+CTG treatment will be performed in all cases. Participants will be assessed at 6 weeks, 3 months, and 6 months to evaluate clinical, volumetric, and patient-centred outcomes.

DETAILED DESCRIPTION:
In this investigation, a prospective cohort study, several key outcomes will be assessed. First, we seek to determine whether restoring the cementoenamel junction (CEJ) in Class B GRs before root coverage therapy yields comparable clinical and volumetric outcomes to Class A GRs with detectable CEJ. In addition, the influence of the CEJ restoration on dentin sensitivity and aesthetic satisfaction of the patient will be investigated. To our knowledge, it will be the first clinical study to use Pini Prato et al.'s surface discrepancy classification as a decision-making tool to guide periodontal-restorative procedures.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals older than 18 years old;
* Healthy periodontal status according to the AAP/EFP definition;
* Full-mouth plaque (FMPS) and bleeding scores (FMBS) ≤ 20%;
* At least one facial RT1 GR in single-rooted teeth with a minimum depth of 2 mm, associated with a NCCL;
* No history of periodontal surgery at the experimental site(s).

Exclusion Criteria:

* Pregnancy or lactation;
* Self-reported smoking ≥10 cigarettes/day;
* Metabolic diseases that negatively affect soft tissue healing (i.e., diabetes mellitus);
* Any medication that may interfere with wound healing;
* Prosthetic crown at experimental teeth;
* Ongoing orthodontic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-26 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Mean Root Coverage (MRC) | 6 months
  Mean root coverage assessed in percentage

SECONDARY OUTCOMES:
Complete Root Coverage (CRC) | 6 months
  Complete Root Coverage assessed in percentage
Change in keratinized tissue width (ΔKTW) | 6 weeks, 3 months, 6 months
  Change in keratinized tissue width assessed digitally in mm
Change in marginal gingival thickness (ΔMGT) | 6 weeks, 3 months, 6 months
  Change in marginal gingival thickness assessed at 1, 2, and 3 mm from the gingival margin in mm
Change in recession depth (ΔRD) | 6 weeks, 3 months, 6 months
  Change in recession depth assessed digitally in mm
Change in recession area (ΔRA) | 6 weeks, 3 months, 6 months
  change in recession area assessed digitally in mm^2
Change in mucosal volume (ΔMV) | 6 weeks, 3 months, 6 months
  change in mucosal volume assessed digitally in mm^3
Probing pocket depth (PPD) | 6 months
  probing pocket depth assessed clinically in mm using a periodontal probe
Clinical attachment level (CAL) | 6 months
  Clinical attachment level assessed clinically in mm (sum of probing pocket depth and recession)
Dentin sensitivity as assessed by VAS (Visual Analog Scale) | Initial, 6 months
  Dentin sensitivity assessed on each tooth after directing an air blast from a triple syringe at the buccal cervical areas, maintaining a distance of 1 cm for 5 seconds, using a Visual Analog Scale [0-100]
Patient aesthetic satisfaction as assessed by VAS (Visual Analog Scale) | 6 months
  Patient aesthetic satisfaction assessed using a Visual Analog Scale [0-100]

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Blasi, Study Director — Universitat Internacional de Catalunya; José Nart, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- BLASI Clínica Dental Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No